CLINICAL TRIAL: NCT02299557
Title: A Double Blind Study to Examine the Effect of Oxymetazoline Gel on Anal Pressure and Incontinence in Spinal Cord Injury Patients
Brief Title: The Effect of Oxymetazoline Gel on Anal Pressure and Incontinence in Spinal Cord Injury Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDD 116
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Fecal Incontinence; Spinal Cord Injury
MeSH Terms: conditions — Fecal Incontinence; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment (Experimental): Intra-anal Oxymetazoline gel once daily
  Interventions: Drug: Oxymetazoline gel
- Placebo (Placebo Comparator): Intra-anal Placebo gel once daily
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Oxymetazoline gel — Oxymetazoline gel applied intra-anally once daily
  Arms: Treatment
Drug: Placebo gel — Placebo gel applied intra-anally once daily
  Arms: Placebo

SUMMARY:
This is an double blinded, cross-over study to determine the effect of Oxymetazoline gel on anal resting pressure and fecal incontinence in patients with spinal cord injury. Approximately 17 subjects are expected to complete this 10 weeks study that will include two treatment periods of 4 weeks each, and one 2 weeks wash out period.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female subjects 18 to 55 years of age;
* Spinal Cord Injury that occurred at least 3 months from randomization day and less than 3 years from randomization day.
* At least 4 unwanted/unexpected incontinent events/week

Exclusion Criteria:

* Known allergy to Oxymetazoline or silicone.
* Pregnancy or lactation.
* Active cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities;
* Type 1 diabetes mellitus;
* Insulin treated type 2 diabetes mellitus;
* Renal insufficiency.
* Liver insufficiency.
* Malignant disease within 5 years of screening;
* History of rectal surgery.
* History of HIV, hepatitis B, hepatitis C.
* Has upon physical examination a rectal deformation or signs of rectal disease such as fissure, bleeding hemorrhoids, fistula, infection or space occupying lesion.
* Has used, in the last 1 week, drugs that may affect blood coagulation, such as Aspirin (at a dose above 500 mg/day), Warfarin, Sintrom, Enoxaparin, Nadroparin, Heparin, Clopidogrel, Ticlopidine.
* Hypertension (blood pressure over 150/105 mm Hg in screening visit)
* Unable to understand the use instruction, as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To examine the effect of Oxymetazoline gel on fecal incontinence episodes in the 8 hours following application. | 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetics (area under the curve [AUC]), peak concentration and half life time (T 1/2) of Oxymetazoline; | 4 weeks
Number of participants with adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis Egyetem I. sz. Belgyógyászati Klinika, Budapest, Hungary